CLINICAL TRIAL: NCT05838469
Title: Clinical Evaluation of High Viscosity Glass Ionomer Strip Crowns in Primary Maxillary Incisors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Beste Ozgur, assistant professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUDHF-StripCrown
Record Dates: First submitted 2023-04-10; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Early Childhood Caries
Keywords: high viscosity glass ionomer cement; strip crown; pediatric dentistry; child; early childhood caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strip Crown (Experimental): This is a single-arm study. High viscosity glass ionomer strip crowns will be performed to all patients.
  Interventions: Other: Pediatric Strip Crown and High Viscosity Glass Ionomer Cement

INTERVENTIONS:
Other: Pediatric Strip Crown and High Viscosity Glass Ionomer Cement — Following the decision on the appropriate size of celluloid strip crown, the tooth will be isolated using roll cottons and the "cavity conditioner" (GC, Japan) will be applied to all surfaces for 10 seconds, washed away and dried with cotton pellets. The selected celluloid strip crown will be filled with a fluoride-releasing bulk fill hybrid glass ionomer cement (EQUIA Forte, GC, Japan) prepared by mixing for 10 seconds in an automatic mixer and placed on the tooth with light pressure. The excess material on the crown margins will be removed with a hand instrument, and the celluloid strip crown will be removed from the tooth. If necessary, the restoration will be polished using a polishing discs. After the crown surface is washed and dried, a nano-filled surface sealant (EQUIA Forte Coat, GC, Tokyo, Japan) will be applied for 10 seconds with a micro-tipped applicator and light cured for 20 seconds.

SUMMARY:
The aim of this study was to evaluate the clinical success of modified celluloid strip crown restorations applied using interim therapeutic restoration and high-viscosity glass ionomer cement to the maxillary anterior teeth of children with early childhood caries and cooperation problems.

DETAILED DESCRIPTION:
Following the decision on the appropriate size of celluloid strip crown, the tooth will be isolated using roll cottons and the "cavity conditioner" (GC, Japan) will be applied to all surfaces for 10 seconds, washed away and dried with cotton pellets. The selected celluloid strip crown will be filled with a fluoride-releasing bulk fill hybrid glass ionomer cement (EQUIA Forte, GC, Japan) prepared by mixing for 10 seconds in an automatic mixer and placed on the tooth with light pressure. The excess material on the crown margins will be removed with a hand instrument, and the celluloid strip crown will be removed from the tooth. If necessary, the restoration will be polished using a polishing discs. After the crown surface is washed and dried, a nano-filled surface sealant (EQUIA Forte Coat, GC, Tokyo, Japan) will be applied for 10 seconds with a micro-tipped applicator and light cured for 20 seconds. Clinical evaluations will be done at the 3rd, 6th and 12th months.

ELIGIBILITY:
Inclusion Criteria:

* Read the informed consent form and agree to participate in the study
* Healthy children, aged 2-6 years
* Presenting at least one primary anterior tooth with a class I, II, IV or V caries lesion

Exclusion Criteria:

* Uncooperative children
* The need for vital or non-vital endodontic treatment in the primary tooth to be treated
* Previously restorated tooth
* Presence of bruxism, Class III occlusion or deep bite

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 12 months regarding "Anatomic form" | baseline, 3-month, 6-month,12-month
  alpha: The general contour of the restorations follows the contour bravo: the general contour of the restoration does not follow the contour of the tooth charlie: The restoration has an overhang does
Change from baseline to 12 months regarding "Marginal adaptation" | baseline, 3-month, 6-month,12-month
  alpha: Explorer does not catch or has one-way catch when drawn across the restoration/tooth interface bravo: explorer falls into crevice drawn across the restoration/tooth interface charlie: Dentin or base is exposed along the margin bravo: The general contour of the restoration does not follow the contour of the tooth charlie: The restoration has an overhang does
Change from baseline to 12 months regarding "Surface roughness" | baseline, 3-month, 6-month,12-month
  alpha: the surface of the restoration does not have any surface defects bravo: the surface of the restoration has minimal surface defects charlie: the surface of the restoration has severe surface defects
Change from baseline to 12 months regarding "Marginal staining" | baseline, 3-month, 6-month,12-month
  alpha: there is no discoloration between the restorations and tooth bravo: there is discoloration on less than half of the circumferential margin charlie: there is discoloration on more than half of the circumferential margin
Change from baseline to 12 months regarding "Retention" | baseline, 3-month, 6-month,12-month
  alpha: intact bravo: chipped/loss of material charlie: complete loss of crown
Change from baseline to 12 months regarding "Incisal wear" | baseline, 3-month, 6-month,12-month
  alpha: intact bravo: wear of occlusal surface without tooth surface exposure charlie: wear of occlusal surface with tooth surface exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waggoner WF. Restoring primary anterior teeth: updated for 2014. Pediatr Dent. 2015 Mar-Apr;37(2):163-70. PMID 25905657
- [Background] Policy on Early Childhood Caries (ECC): Unique Challenges and Treatment Options. Pediatr Dent. 2016 Oct;38(6):55-56. No abstract available. PMID 27931421
- [Background] Policy on Interim Therapeutic Restorations (ITR). Pediatr Dent. 2018 Oct 15;40(6):58-59. No abstract available. PMID 32074851
- [Background] Friedl K, Hiller KA, Friedl KH. Clinical performance of a new glass ionomer based restoration system: a retrospective cohort study. Dent Mater. 2011 Oct;27(10):1031-7. doi: 10.1016/j.dental.2011.07.004. Epub 2011 Aug 15. PMID 21840585